CLINICAL TRIAL: NCT05475132
Title: Effects of Exergaming on Bimanual Hand Dexterity in Autistic Children
Brief Title: Exergaming on Hand Dexterity In Autistic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/22/0204 Maham Shabbir
Record Dates: First submitted 2022-07-14; First posted 2022-07-26 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Exergaming; Dexterity
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Exergaming

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergaming (Experimental): App based exercise games for dexterity will be used
  Interventions: Other: Exergaming
- Conventional Dexterity Exercises (Active Comparator): Dexterity exercises used conventionally will be done in this.
  Interventions: Other: Conventional Dexterity Exercises

INTERVENTIONS:
Other: Exergaming — exercise games will be done for a total of 8 weeks ,100min of exergaming/week (5 days × 20 min).
  Arms: Exergaming
Other: Conventional Dexterity Exercises — Exercises traditionally used for dexterity will be done for 8 weeks, 100min of exercises/week (5days × 20 min)
  Arms: Conventional Dexterity Exercises

SUMMARY:
Through this study we aim to determine the effect of Exergaming on bimanual hand dexterity in Autistic children. This randomized controlled trial will recruit a sample of 20 autistic children as per the inclusion and exclusion criteria, through convenient sampling. The sample will be then randomly allocated to control group receiving the conventional dexterity training exercises and Intervention group which will be receiving conventional plus exergaming intervention.

DETAILED DESCRIPTION:
A study showed that a structured traditional physical activity intervention that targets specific MS resulted in motor function improvement in children with ASD along with exergaming that can improve EF in children with ASD.

On a population of 20 patients with CP, Structured Neurodevelopmental Therapy-based hand rehabilitation (SNDTBHR) was applied and in the results Positive effects of both interventions i.e. SNDTBHR and LMBET were found. Significant differences were found between LMBET and SNDTBHR on GGF, pinch forces, JHFT, and WCST all being in the favor of LMBET. Exergaming interventions in the individuals with ASD showed significant improvements in the physical fitness, executive functioning, and their self perception. Exergaming increased the interest and participation of Autistic children in moderate-to-vigorous physical activity. In contrast, exergaming had small impact on emotional regulation As per the results of another study participants with poorer dexterity in the beginning of exergaming training program greatly improved their dexterity performance, which also improved their quality of life. Adherence and motivation increased significantly and system usability of the exergaming was acceptable. Participants with impaired dexterity showed improvement in the Nine-Hole Peg Test and the PDQ-39

According the researchers knowledge there have been numerous studies conducted on the effect of different exercise protocols on autistic children but there is lack of evidence in determining the effect of exergaming on specifically hand functioning/ dexterity in autistic population'. More studies should be done in order to check if exergaming or conventional treatment differ in their effect on hand dexterity in autistic children. Home based exergaming and low cost video assisted games for dexterity need more in depth study so that they can be readily used by general public.

ELIGIBILITY:
INCLUSION CRITERIA:

* Male and female children pre-diagnosed with autism spectrum disorder.
* Autistic Children who are compliant with exergaming

EXCLUSION CRITERIA

* Children not pre-diagnosed with autism spectrum disorder
* Autistic Children who have other coordination disorder such as developmental coordination disorder
* Autistic Children with upper limb amputation.
* Autistic children with loss of vision

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Minnesota Manual Dexterity Test (MMDT) | 4 weeks
  This test evaluates the gross motor skill of the assessed individual, including the the unilateral and bilateral manual dexterity. It is used for various purposes including the measurement of disability , specific training programs and manual activities in practical life, as to hand grip strength

SECONDARY OUTCOMES:
Box and Block Tests (BBT) | 4 weeks
  It is designed to measure manual dexterity, which often underestimated in assessment of patients. The BBT consists of transporting small pieces of wood from one side to the other for one minute. These blocks must be taken from end to end from a wooden box with partition. The number of blocks has to be recorded for the upper dominant and non-dominant member upon three attempts for each member

CONTACTS AND LOCATIONS:
Overall Officials: Sara Aabroo, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - CARD(Clinic for autism and related disorders), Lahore, Punjab Province
  - Lahore Autism Centre, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lord C, Brugha TS, Charman T, Cusack J, Dumas G, Frazier T, Jones EJH, Jones RM, Pickles A, State MW, Taylor JL, Veenstra-VanderWeele J. Autism spectrum disorder. Nat Rev Dis Primers. 2020 Jan 16;6(1):5. doi: 10.1038/s41572-019-0138-4. PMID 31949163
- [Background] Kim SK. Recent update of autism spectrum disorders. Korean J Pediatr. 2015 Jan;58(1):8-14. doi: 10.3345/kjp.2015.58.1.8. Epub 2015 Jan 31. PMID 25729393
- [Background] Paquet A, Olliac B, Golse B, Vaivre-Douret L. Nature of motor impairments in autism spectrum disorder: A comparison with developmental coordination disorder. J Clin Exp Neuropsychol. 2019 Feb;41(1):1-14. doi: 10.1080/13803395.2018.1483486. Epub 2018 Jun 20. PMID 29923455
- [Background] Pixa NH, Steinberg F, Doppelmayr M. High-definition transcranial direct current stimulation to both primary motor cortices improves unimanual and bimanual dexterity. Neurosci Lett. 2017 Mar 16;643:84-88. doi: 10.1016/j.neulet.2017.02.033. Epub 2017 Feb 14. PMID 28229937
- [Background] Fulceri F, Grossi E, Contaldo A, Narzisi A, Apicella F, Parrini I, Tancredi R, Calderoni S, Muratori F. Motor Skills as Moderators of Core Symptoms in Autism Spectrum Disorders: Preliminary Data From an Exploratory Analysis With Artificial Neural Networks. Front Psychol. 2019 Jan 9;9:2683. doi: 10.3389/fpsyg.2018.02683. eCollection 2018. PMID 30687159
- [Background] Friel KM, Kuo HC, Fuller J, Ferre CL, Brandao M, Carmel JB, Bleyenheuft Y, Gowatsky JL, Stanford AD, Rowny SB, Luber B, Bassi B, Murphy DL, Lisanby SH, Gordon AM. Skilled Bimanual Training Drives Motor Cortex Plasticity in Children With Unilateral Cerebral Palsy. Neurorehabil Neural Repair. 2016 Oct;30(9):834-44. doi: 10.1177/1545968315625838. Epub 2016 Feb 11. PMID 26867559
- [Background] Fang Q, Aiken CA, Fang C, Pan Z. Effects of Exergaming on Physical and Cognitive Functions in Individuals with Autism Spectrum Disorder: A Systematic Review. Games Health J. 2019 Apr;8(2):74-84. doi: 10.1089/g4h.2018.0032. Epub 2018 Oct 17. PMID 30332294
- [Background] Rafiei Milajerdi H, Sheikh M, Najafabadi MG, Saghaei B, Naghdi N, Dewey D. The Effects of Physical Activity and Exergaming on Motor Skills and Executive Functions in Children with Autism Spectrum Disorder. Games Health J. 2021 Feb;10(1):33-42. doi: 10.1089/g4h.2019.0180. Epub 2020 Dec 23. PMID 33370161
- [Background] van Beek JJW, van Wegen EEH, Bohlhalter S, Vanbellingen T. Exergaming-Based Dexterity Training in Persons With Parkinson Disease: A Pilot Feasibility Study. J Neurol Phys Ther. 2019 Jul;43(3):168-174. doi: 10.1097/NPT.0000000000000278. PMID 31136450
- [Background] Gao Z, Zeng N, Pope ZC, Wang R, Yu F. Effects of exergaming on motor skill competence, perceived competence, and physical activity in preschool children. J Sport Health Sci. 2019 Mar;8(2):106-113. doi: 10.1016/j.jshs.2018.12.001. Epub 2018 Dec 6. PMID 30997256